CLINICAL TRIAL: NCT06665620
Title: BRITE 2.0: A Just-in-time Adaptive Intervention for Suicide Safety Planning in Adolescents
Brief Title: Optimizing a Just-in-time Adaptive Intervention for Suicide Safety Planning in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ksana Health (Industry)
Collaborators: University of Pittsburgh Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OV-003; R44MH135605 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Mental Health Disorder; Anhedonia
Keywords: depression; depressive disorder; mood disorder; mental disorders; suicidal behaviors; suicidal thoughts; suicidal ideation
MeSH Terms: conditions — Suicide; Mental Disorders; Anhedonia; Depression; Depressive Disorder; Mood Disorders; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: At each decision point (once per day), participants will be randomized to receive a n nudge encouraging them to access the ViraBrite app and utilize suicide safety planning skills vs. no nudge. At each decision point, participants will have a seventy-five percent chance of receiving a nudge. Given that they are randomized to receive a nudge, participants have a 33.3% chance of receiving a notification at one of three time points: morning, midday or evening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ViraBrite (Experimental): Each day, participants will receive nudges according to a micro-randomized pattern that encourage them to access the ViraBrite app and utilize coping and suicide safety planning skills. One decision point will occur per day. At each decision point, participants will have a seventy-five percent chance of receiving a nudge. Given that they are randomized to receive a nudge, participants have a 33.3% chance of receiving a notification at one of three time points: morning, midday or evening.
  Interventions: Behavioral: ViraBrite nudges

INTERVENTIONS:
Behavioral: ViraBrite nudges — Each day, participants will receive prompts via smartphone notifications that encourage them to access the ViraBrite app and utilize suicide safety planning skills.

SUMMARY:
Despite efforts to prevent suicide, US rates are climbing, and suicide is the second leading cause of death amongst youth. Digital tools, especially personal smartphones, are promising avenues to address these issues and can be used to increase engagement with effective interventions such as suicide safety planning. The BRITE suicide safety planning app was developed on evidence-based principles and has undergone rigorous formative development and effectiveness evaluations. However, to optimize its functionality, commercial viability, and scale its implementation, issues related to user engagement need to be addressed. This 4-week Micro-Randomized Trial (MRT) will optimize specific components of ViraBrite, an augmented version of the BRITE suicide safety planning app that integrates automated algorithms (i.e., just in time adaptive intervention features) to facilitate increased engagement with coping skills and pushes safety planning materials to users at periods of high risk (i.e., increases in emotional distress).

DETAILED DESCRIPTION:
The goal of the MRT is to optimize the ViraBrite intervention by randomly assigning participants to various combination of notification timing (e.g., morning, midday, evening). Participants will download the ViraBrite suicide safety planning app that integrates automated algorithms (i.e., just in time adaptive intervention features) to facilitate increased engagement with coping skills and pushes safety planning materials to users at periods of high risk (i.e., increases in emotional distress). The MRT will last for 4 weeks for each participant. Each day, participants will receive prompts ("nudges") according to a micro-randomized pattern that encourage them to access the ViraBrite app and utilize suicide safety planning skills. One decision point will occur per day. At each decision point, participants will have a seventy-five percent chance of receiving a nudge. Given that they are randomized to receive a nudge, participants have a 33.3% chance of receiving a notification at one of three time points: morning, midday or evening. The MRT will also investigate the impact of estimated emotional distress as a moderator of responding to the nudge. Specifically, measures of distress including 1. Self-report of daily mood, 2. Linguistic markers of distress (i.e., first person pronoun use) and 3. Geolocation will be explored as moderators of engagement with nudges.

ELIGIBILITY:
Inclusion Criteria:

* Recent suicide attempt or ideation with a plan
* English fluency and literacy
* Parent or legal guardian willing and able to legally provide informed consent

Exclusion Criteria:

* Unable to read/understand English
* Current manic or psychotic episode
* Development disability precluding comprehension of study procedures
* No routine access to a mobile phone, assessed by EHR review and during phone screen
* No eligible parent or legal guardian to provide informed consent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Proximal engagement with ViraBrite | 24 hours
  Engagement with the ViraBrite app (i.e., tapping on the push notification, patterns of accessing app features such as coping skills and safety plan) between the current and next randomization
Engagement with ViraBrite | 4 weeks
  Engagement over the course of the trial will be measured through objective app usage metrics, including total number and frequency of features used

SECONDARY OUTCOMES:
Mood and Feelings Questionnaire (MFQ) | 4 weeks
  The MFQ is a 13-item self-report questionnaire used to screen for depressive in children and young people. Items are rated on a 3-point Likert scale (not true = 0; sometimes true = 1; not true = 2). Scores are calculated by summing the point values on each response. Total MFQ scores range from 0 to 26, with higher scores suggesting greater severity in depressive symptoms.
Snaith-Hamilton Pleasure Scale (SHAPS) | 4 weeks
  The SHAPS is a 14-item scale that measures anhedonia. The items cover the domains of social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Thus, the final score ranges from 0 to 14. Higher scores indicate greater anhedonia.
Screen for Anxiety Related Emotional Disorders (SCARED) | 4 weeks
  The SCARED is a 5-item self-report questionnaire used to screen for childhood anxiety disorders including general anxiety disorder, separate anxiety disorder, panic disorder, and social phobia. Items are rated on a 3-point Likert scale from 0 to 2 and summed to yield a total score. Total scores range from 0 to 10. Higher scores indicate greater anxiety.
Reasons for Living | 4 weeks
  The Reasons for Living (RFL) Inventory is a 48-item instrument that measures a range of beliefs potentially important as reasons for not committing suicide. The items are rated on 6-point Likert type scales based on how important each reason would be for living if suicide was contemplated (1 = not at all important; 6 = extremely important). The total score is calculating by calculating the mean of the item scores and multiplying the result by 48. Total scores can only be calculated if a participant answers at least 38 items.
Columbia Suicide Severity Rating Scale (C-SSRS) | Weekly
  The C-SSRS is an assessment of suicidal thoughts and behaviors in clinical and research settings. The C-SSRS consists of 16 questions about suicidal thoughts and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). This 5-item subscale ranges from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States